CLINICAL TRIAL: NCT03612310
Title: Developing Protocols for Modelling of Genetic Diseases Using Induced Pluripotent Stem Cells
Status: Not yet recruiting | Type: Observational
Sponsor: Kevin Bruce (Industry)
Responsible Party: Sponsor-Investigator, Kevin Bruce, Chief Operating Officer, Censo Biotechnologies Ltd
Organization: Censo Biotechnologies Ltd (Industry)
Other Study IDs: 18/SS/0061
Record Dates: First submitted 2018-06-15; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Cell lines derived from skin, urine or blood. No primary tissue retained. All samples anonymised. All samples consented for genetic analysis of cultured cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Skin biopsy/Urine Collection/Blood Sample Collection — Participant will meet clinician in a suitable local clinical setting, in select circumstances the clinician may attend the participants home. Clinician will collect a 5-7mm section of skin, the area may be numbed beforehand and stitches may be used to close the wound when required. The wound will be dressed if deemed necessary by medical professional.
  Participant will meet clinician in a suitable local clinical setting, in select circumstances the clinician may attend the participants home. The clinician or phlebotomost will use a disposable needle to remove a blood sample (normally 50ml but could be up to 320ml for adults).
  Participant will meet clinician in a suitable local clinical setting, in select circumstances the clinician may attend the participants home. The clinician or other nominated member of the clinical team will provide a sterile urine collection vessel and direct the volunteer to a suitable private toilet area to provide the sample.

SUMMARY:
Recent advances have shown that cells from human blood, skin and urine samples can be reprogrammed to become stem cells. These are called induced Pluripotent Stem Cells (iPSCs) and share many characteristics with embryonic stem cells, including an unlimited capacity for proliferation and the potential to become any cell in the body. Beneficially, the use of iPSCs avoids the ethical difficulties which surround embryonic stem cells and allows generation of iPSC lines which are disease representative. For example, we could take skin samples from an individual diagnosed with Huntington's disease and their unaffected sibling and using this technology, generate iPSC lines from both individuals. Using these iPSCs, we could produce disease affected cell populations from the affected and unaffected individuals, use these cells to research why specific cell populations are affected by disease and test new treatments to combat disease progression, essentially producing a 'disease in a dish'. This is just one example of many for which this technology could be applied. We can also utilise gene-editing techniques to generate isogenic controls or insert disease related mutations to assess disease phenotype.

Although generation of iPSC lines has been robustly proven across multiple disease backgrounds, many aspects of their downstream use still remain to be determined. Particularly, robust protocols for directing iPSCs towards cell fates such as neurons or blood cells must be developed to fully realise application of iPSCs in disease modelling and drug screening.

This study involves the collection of human blood, skin or urine samples from subjects bearing a range of genetic diseases alongside those from individuals who have not been diagnosed with a disease, as controls. These samples will be used to generate iPSC lines for development of differentiation and disease phenotyping protocols.

DETAILED DESCRIPTION:
Recent advances in biotechnology have shown that somatic cells (such as skin, blood and urine cells) from human adults and children can be reprogrammed to change their characteristics and become other types of cells that may be useful for disease modelling and drug screening. This includes the generation of induced pluripotent stem cells (iPS cells) which can be derived from these somatic cells by a process known as "cellular reprogramming". These iPSCs share many characteristics with embryonic stem cells, including an unlimited capacity for proliferation and the potential to differentiate into any cell of the body. However, unlike embryonic stem cells, the generation of iPSCs avoids the practical and ethical difficulties of obtaining embryonic tissues. Consequently, cellular reprogramming and iPSC technology has great implications in the field of disease modelling and drug screening.

Many obstacles must be overcome before iPSC based disease modelling and drug screening can fully be realised and allow replacement of inadequate animal models and simplistic cell models. This study will enable us to gather samples from a range of participants from different disease backgrounds, and to develop suitable panels of iPSCs for the purpose of protocol development. Development of robust protocols which are suitable for use across multiple iPSC lines and repeatable across multiple laboratories are essential for the use of iPSCs in disease modelling and drug screening. This study will allow us to look at causation of disease across a range of disease specific cell lines with known genetic backgrounds which are representative of a cohort of human patients. This is fundamental for development of iPSC based drug screening assays.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Individuals diagnosed with a genetic disease - any age between 1-120 years.
* Individuals diagnosed with a genetic disease - must be able to communicate well with the investigator and to comply with the requirements of the entire study OR be under the care of an appropriate guardian, if incapacitated or under the age of 16.
* Individuals diagnosed with a genetic disease - require provision of written informed consent either by participant or guardian, to participate as shown by a witnessed signature on the Subject Consent Form
* Individuals participating as controls - aged between 16-120 years.
* Individuals participating as controls -must be able to consent for themselves

Exclusion Criteria:

* Individuals less than 1 year old.
* Infection with any blood borne diseases (e.g. HIV, Hepatitis B or Hepatitis C).
* Previous or current intravenous drug abuse.
* For donation of blood samples only - has exceeded annual limit for blood donation.
* Affected by blood disorders such as anaemia, blood clotting disorders or currently on anticoagulant drug therapy.
* Individuals participating as controls - excluded if aged less than 16 years old.
* Individuals participating as controls - excluded if unable to consent for themselves.
* Individuals diagnosed with a genetic disease - unable to provide informed consent either by themselves or through an appropriate nearest relative, legal guardian or welfare attorney.

Ages: 1 Year to 120 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with genetic diseases and/or healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of disease relevant iPSC differentiation protocols generated within the study | 2 years
  The primary research question is to determine if and how we can use iPSCs to improve modelling of genetic diseases, particularly in generating iPSC-derived, disease relevant, tissue specific cell populations. Currently, research into the pathology and progression of genetic diseases and subsequent development of therapeutics is heavily dependent on the use of simplistic cell models and/or animal models which are poorly representative of the human disease. Although generation of iPSC lines has been observed across many disease backgrounds, a number of facets of their downstream use still remain to be determined. To fully exploit the possibilities of iPSCs, it is critical to develop differentiation protocols (that is, directing iPSCs to form populations of other cell types, such as neurons or cardiomyocytes) which are robust and reliable across multiple cell lines when performed in a high throughput manner.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Bruce, BSc, Study Director — Censo Biotechnologies Ltd

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymised / anonymised data will be disseminated via peer reviewed scientific journals, internal reports and scientific presentations.

REFERENCES:
- See also: Censo Biotechnologies Website — http://www.censobio.com